CLINICAL TRIAL: NCT05696314
Title: Surgeon-performed Outpatient Transoral and Transcervical Ultrasound Compared to MRI for the Diagnostic Workup of Primary Oropharynx Tumors: the SPOT-US Trial
Brief Title: Surgeon-performed Outpatient Transoral and Transcervical Ultrasound of the Oropharynx
Acronym: SPOT-US
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Martin Garset-Zamani, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Transoral Ultrasound
Record Dates: First submitted 2022-12-16; First posted 2023-01-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-08

CONDITIONS: Oropharynx Cancer; Tonsil Cancer; Base of the Tongue Tumor; Tonsil Hypertrophy; Tonsil Ulcer; Tonsil Neoplasm; Tonsil Lymphoma; Base of Tongue Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Tonsillar Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention (transoral and transcervical ultrasound) is performed on all included patients. All patients will also receive a standard MRI of the oropharynx. All tumors will be biopsy verified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Outpatient Oropharynx Ultrasound (Experimental): Transoral and/or Transcervical ultrasound of the oropharynx
  Interventions: Diagnostic Test: Transoral Ultrasound; Diagnostic Test: Transcervical Ultrasound

INTERVENTIONS:
Diagnostic Test: Transoral Ultrasound — The oropharynx is scanned using high-frequency, small-footprint ultrasound transducers placed onto the suspected oropharynx sub-locations (e.g. tonsils or tongue base). Lidocaine spray or gel will be applied prior to scanning to reduce the gag reflex.
Diagnostic Test: Transcervical Ultrasound — Curved low-frequency ultrasound transducers will be placed on the submental region on the skin of the neck, and the tongue base will be visualized in the midline in transverse and sagittal planes. The tonsils will be visualized adjacent to the tongue base on either side in oblique transverse and oblique sagittal planes, deep to the submandibular glands.

SUMMARY:
The purpose of the study is to compare the sensitivity and specificity of transoral ultrasound, transcervical ultrasound, Magnetic Resonance Imaging (MRI) and Positron Emission Tomography-Computerized Tomography (PET-CT) in terms of detecting primary oropharynx tumors.

DETAILED DESCRIPTION:
A prospective study will be performed at the head & neck departments at Copenhagen University Hospital - Rigshospitalet, Zealand University Hospital - Køge, and Aarhus University Hospital in Denmark.

Patients referred with a suspected cancerous lesion of the oropharynx will be invited to participate in this study. With written informed consent, a surgeon-performed outpatient transoral and transcervical examination of the tonsils and tongue base is conducted as an addition to the clinical workup at the head & neck departments. Clinical work-up includes palpation of the oropharynx, flexible endoscopic exam with narrow-band imaging and neck ultrasound.

Ultrasound of the oropharynx will be performed using small-footprint, high-frequency (minimum 15MHz) transducers for transoral ultrasound. A lower-frequency (between 2-9 MHz) curved transducer will be used for transcervical ultrasound. If a suspected tumor is visualized, the location is noted and the surgeon performing clinical examination is informed.

MRIs will be performed on all patients with cancers, and an expert radiologist blinded to ultrasound results will assess all images for tumor detection, greatest tumor size and T-stage. PET/CTs will be performed in patients with suspected cancer of unknown primary tumor as well as patients with verified cancers. A nuclear medicine physician and an oncoradiologist will separately assess PET/CTs and CTs for tumor detection.

Surgeons performing initial clinical work-up, the ultrasound operators, neuroradiologist and nuclear medicine physician will register tumor detection (sub-location specific) and greatest tumor size immediately and prospectively, blinded to histopathology. Prospective gathered data will be registered on standardized data collection sheets or in REDCap using the same standardized variables. All scanning modalities will be evaluated blinded to each other but not to clinical findings.

Tumor detection: Suspected tumor locations from clinical evaluation with narrowband imaging and palpation, ultrasound, MRI, and PET-CT will be categorized according to the following criteria:

* Right tonsil
* Left tonsil
* Right tongue base
* Left tongue base
* Right overlapping tonsil and tongue base
* Left overlapping tonsil and tongue base
* Other oropharynx (soft palate, uvula, anterior and posterior pharyngeal arches, posterior oropharynx wall, and vallecula)
* Multiple tumor locations The examiners' tumor suspicion confidence will be rated with a 5-point Likert scale ranging from 0, very low suspicion - 5, very high suspicion.

The surgeon will also mark on a pictogram of the oropharynx with the biopsy location(s) numbered according to the histopathology registered biopsy locations.

Tumor size and staging: If a tumor is visualized or palpated, the greatest tumor diameter will be measured in three dimensions with clinical palpation, ultrasound, and MRI. T-staging will be estimated according to the Union for International Cancer Control 8th edition TNM-staging system:

* Tx: Unknown primary tumor.
* T1: Tumor <20 mm in greatest diameter.
* T2: Tumor 21-40 mm in greatest diameter.
* T3: Greatest size >40mm or extension to the lingual surface of the epiglottis
* T4: Invasion of the extrinsic tongue muscles, larynx, pterygoid muscles, hard palate, mandible, carotids nasopharynx or skull base (yes, no, indeterminate).

Additional variables: We will prospectively register the study center, date of outpatient ultrasound, ultrasound machine used, doctor performing the ultrasound scan, patient Mallampati 4-point score, Patient mouth opening measured in millimeters between incisors, patient self-reported discomfort from transoral ultrasound and palpation examinations (Supplementary Figure 2), ultrasound scan quality, MRI scan quality and PET-CT scan quality. Quality will be registered on a 5-point Likert scale (1, Very poor quality - 5, excellent quality).

The following data will be registered from medical charts: patient age, sex, tobacco smoking, alcohol consumption, date of first clinical contact, date of MRI scan performed, date of PET/CT scan performed, date of available histopathology results and date of treatment initiation.

Ultrasound video clips and B-mode images will be stored for retrospective descriptive evaluation of the following characteristics:

* Tumor shape (smooth/rounded, irregular/lobular).
* Tumor border delineation (well-circumscribed, unclear).
* Tumor heterogeneity (homogeneous, heterogeneous).
* Doppler flow compared to contralateral side (decreased, equivocal, increased).
* Doppler flow characteristics (peripheral/circumferential, internal organized, internal chaotic)

Reference standard: Final histopathology biopsy results will define the presence of cancer as binary results (no cancer vs. cancer present). An expert head and neck pathologist will re-evaluate biopsies results if inconclusive. The presence of a tumor in a correct sub-location assessed by final Multidisciplinary Team (MDT) conference will be used to define correct tumor location. Greatest tumor size and T-stage will also be determined by final MDT decision, considering the clinical and radiological findings. For patients with available complete tumor resections, a secondary analysis will be performed using the histopathologic reported greatest tumor diameter as reference standard.

ELIGIBILITY:
Inclusion criteria:

* Initially assessed by a specialist otorhinolaryngologist with clinical suspicion of head and neck cancer and referred to fast-track cancer work-up.
* Any of the following objective or subjective symptoms:

  1. Visible and/or palpable tumors of the oropharynx.
  2. Asymmetry of the tonsils or tongue base.
  3. Symptoms including dysphagia, throat pain, and/or referred otalgia where an oropharynx tumor is suspected but not clinically visible.
  4. Suspected cervical lymph node metastasis with no visible/palpable primary tumor.
  5. Lateral neck cysts in patients aged 40+ years.
* Adult patients aged 18+ years.
* Understands Danish or English and can give written informed consent.

Exclusion criteria:

* Prior radiotherapy to the oropharynx.
* Prior oropharynx cancer.
* MRI of the oropharynx or PET-CT already performed 3 months prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Tumors detected by clinical evaluation, ultrasound, MRI, CT, and PET/CT compared to the reference standard histopathology results. | 2 weeks.
  Sub-location specific detection of tumors in the oropharynx will be assessed blinded to histopathology. The final histopathology diagnosis will typically be available within two weeks.

SECONDARY OUTCOMES:
Greatest tumor diameter in millimeters estimated with clinical evaluation, ultrasound and MRI, and CT. | 1 minute
  The greatest tumor diameter is measured in millimeters.
Categorical T-stage estimated with clinical evaluation, ultrasound, and MRI, and CT. | 1 minute
  Categorized according to the Union for International Cancer Control 8th edition TNM-staging system. Tumors will be categorized double-blinded between ultrasound and MRI.
Tonsil and tongue base tumor volume estimated with clinical evaluation, ultrasound and MRI, and CT. | 1 minute
  Volume is calculated from three perpendicular greatest tumor diameters if available. The volume formula for an ellipse is used: 3/4 * pi * (height/2) * (width/2) * (length/2).

OTHER OUTCOMES:
Comparison of tumor detection and size between MRI and CT | 1 year
  Two radialogists blinded to eachother will retrospectively evaluate tumor detection and greatest tumor size in millimeters on clinically acquired MRI and CT images blinded to histopathology results and tumor measurements.
MRI and PET-CT scan quality | 1 year
  5-point Likert scales for border delineation, internal details and overall quality in tumor suspected tonsils and tongue base will be assessed for each scan.
Ultrasound scan quality | 1 minute
  5-point Likert scales for border delineation, internal details and overall quality in tumor suspected tonsils and tongue base will be assessed for transoral and Transcervical ultrasound at the time the scan is performed.
Patient mouth opening in millimeters. | 1 minute
  The mouth opening in patients is measuredbetween the incisors using a ruler.
11-point Numeric Rating Scale for Discomfort of oropharynx palpation and transoral ultrasound | 1 minute
  Palpation and transoral ultrasound of tonsils and the tongue base will be rated by the patient on a scale from 0, no discomfort, to 10, worst discomfort imaginable.
Gagging severity index | 1 minute
  Patients gagging severity will be rated by the clinical examiner on a 5-point scale (1 - normal gagging, 5 - very severe gagging).
Patient Mallampati score | 1 minute
  The Mallampati score from class I to class IV is evaluated by the surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Todsen, MD, PhD, Study Director — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Århus University Hospital, Department of Otorhinolaryngology, Head & Neck Surgery, Aarhus
  - Rigshospitalet, Department of Otorhinolaryngology, Head & Neck Surgery & Audiology, Copenhagen
  - Zealand University Hospital - Køge, Department of Otorhinolaryngology, Head and Neck Surgery, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garset-Zamani M, Norling R, Hahn CH, Agander TK, von Buchwald C, Todsen T. Transoral Ultrasound in the Outpatient Clinic for the Diagnostic Work-Up of Oropharyngeal Cancer: A Feasibility Study. Cancers (Basel). 2023 Nov 4;15(21):5292. doi: 10.3390/cancers15215292. PMID 37958465